CLINICAL TRIAL: NCT02302872
Title: Mitral Valve Repair Clinical Trial (MAVERIC Trial)
Brief Title: Treatment of Heart Failure and Associated Functional Mitral Valve Regurgitation
Acronym: MAVERIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mvrx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EU010513, AU220816
Record Dates: First submitted 2014-11-18; First posted 2014-11-27 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Mitral Valve Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ARTO system (Experimental)
  Interventions: Device: ARTO System

INTERVENTIONS:
Device: ARTO System

SUMMARY:
The objective of the study is to evaluate the safety and performance of the ARTO System in patients with mitral valve regurgitation (MR) associated with congestive heart failure (CHF).

ELIGIBILITY:
Inclusion Criteria:

1. Is ambulatory, able and willing to comply with the study protocol and has provided written informed consent
2. Age ≥ 18
3. Trans-septal catheterization is determined to be feasible by the treating physician
4. NYHA class II-IV heart failure of any etiology
5. Symptomatic with MR grade ≥ 2+
6. LVEF ≥20% ≤ 50%
7. LVEDD > 50 mm and ≤ 70 mm
8. No anticipated change in patient's cardiac medication regimen anticipated throughout the course of the study.
9. • In the opinion of the investigator and heart surgery team, the patient is not a candidate for surgery, and the use of the ARTO™ System is technically feasible.

Exclusion Criteria:

1. In the opinion of the Investigator, the femoral vein and internal jugular vein cannot accommodate a 16 F catheter or the presence of an inferior vena cava (IVC) filter would interfere with advancement of the catheter or ipsilateral DVT is present
2. Significant structural abnormality of the mitral valve (e.g., flail, prolapse, leaflet calcification)
3. Significant mitral annular calcification
4. Hemodynamic instability (systolic pressure < 90 mmHg without afterload reduction or cardiogenic shock or the need for inotropic support or intra-aortic balloon pump)
5. Prior mitral valve surgery or valvuloplasty or any currently implanted prosthetic valve or VAD
6. History of, or active, rheumatic heart disease
7. History of Atrial Septal Defects (ASD), whether repaired or not
8. History of previously repaired PFO or PFO associated with clinical symptoms (e.g., cerebral ischemia) within 6 months of the planned investigational procedure
9. In the opinion of the investigator, an atrial septal aneurysm is present that may interfere with transseptal crossing
10. Biventricular pacing initiated or anticipated within 6 months of the planned investigational procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-10; Primary Completion 2021-07 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Event Rate to 30 Days post-procedure | <=30 days post procedure
  Major Adverse Events defined as: death, myocardial infarction, cardiac tamponade, device related cardiac surgery, stroke, renal failure
Mitral regurgitation grade and change from baseline to 30 days | <=30 days post procedure
Device Technical Success | procedural
  At exit from cath lab, alive, with Successful access, delivery and retrieval of the device delivery system, and Deployment and correct positioning (including repositioning/recapture if needed) of the single intended device, and No need for additional unplanned or emergency surgery or re-intervention related to the device or access procedure

CONTACTS AND LOCATIONS:
Overall Officials: Andrejs Erglis, MD, Principal Investigator — Pauls Stradins Clinical University Hospital
Locations (9):
- Australia (4):
  - The Wesley Hospital, Auchenflower, Queensland
  - St Andrews Hospital, Adelaide, South Australia
  - Warringal Private Hospital, Heidelberg
  - The Mount Hospital, Perth
- ICPS, Massy, France
- IRCCS San Donato, Milan, Italy
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- United Kingdom (2):
  - Brighton and Sussex University Hospitals, Brighton
  - St Thomas' Hospital, London

REFERENCES:
- [Derived] Erglis A, Narbute I, Poupineau M, Hovasse T, Kamzola G, Zvaigzne L, Erglis M, Erglis K, Greene S, Rogers JH. Treatment of Secondary Mitral Regurgitation in Chronic Heart Failure. J Am Coll Cardiol. 2017 Dec 5;70(22):2834-2835. doi: 10.1016/j.jacc.2017.09.1110. No abstract available. PMID 29191334
- [Derived] Rogers JH, Thomas M, Morice MC, Narbute I, Zabunova M, Hovasse T, Poupineau M, Rudzitis A, Kamzola G, Zvaigzne L, Greene S, Erglis A. Treatment of Heart Failure With Associated Functional Mitral Regurgitation Using the ARTO System: Initial Results of the First-in-Human MAVERIC Trial (Mitral Valve Repair Clinical Trial). JACC Cardiovasc Interv. 2015 Jul;8(8):1095-1104. doi: 10.1016/j.jcin.2015.04.012. Epub 2015 Jun 24. PMID 26117461